CLINICAL TRIAL: NCT06080958
Title: Negative Pressure Wound Therapy in Flap Enhancement
Brief Title: The Negative Pressure Wound Therapy in Flap Enhancement: Clinical Evaluation Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aswan University Hospital (Other)
Responsible Party: Principal Investigator, Ahmed Salah Eldin, principal investigator, Aswan University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Aswan University Hospital
Record Dates: First submitted 2023-10-08; First posted 2023-10-12 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Surgical Flap; Negative-Pressure Dressings

STUDY DESIGN:
Intervention Model Description: Negative pressure wound therapy (vacuum-assisted wound closure) for postoperative flap care
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- High negative pressure group (Active Comparator): A high negative pressure amplitude, (75- 125 mmHg) on continuous mode, is applied over the flaps
  Interventions: Device: NPWT
- Low negative pressure group (Active Comparator): A low negative pressure amplitude, (50- <75 mmHg) on intermittent mode, is applied over the flaps
  Interventions: Device: NPWT
- Control group (Placebo Comparator): Conventional dressing is applied over the flaps
  Interventions: Other: Conventional dressing

INTERVENTIONS:
Device: NPWT — the NPWT dressing applied to fasciocutaneous flap
  Other Names: VAC
  Arms: High negative pressure group; Low negative pressure group
Other: Conventional dressing — Conventional dressing ( topical care ) applied to fasciocutaneous flap
  Arms: Control group

SUMMARY:
The goal of this study is to compare the clinical outcomes of using NPWT dressing versus conventional dressing in improving flaps outcome

DETAILED DESCRIPTION:
The cases will be divided into 3 major study groups:

1st group will be managed with high negative pressure wound therapy The 2nd group will be managed with low negative pressure wound therapy The 3rd group will be managed with conventional dressing

ELIGIBILITY:
Inclusion Criteria:

- Adult patients skin and soft tissue defects that need flap coverage

Exclusion Criteria:

* associated severe regional injuries uncontrolled comorbidities

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 65 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Number of Participants with primary healing | 2 weeks
  Healing by epithelization without the need for secondary intervention

SECONDARY OUTCOMES:
Number of Participants with flap Edema | 1 week
  flap edema clinical & radiological assessment
Number of Participants with flap Congestion | 1 week
  flap congestion clinical assessment
Number of Participants with flap Ischemia | 1 week
  flap ischemia clinical assessment
Number of Participants with flap infection | 2 weeks
  surgical site infection

CONTACTS AND LOCATIONS:
Locations (1):
- Aswan University Hospital, Aswān, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Elbanna OH, Eldine AS, Sayed AM, Mousa AK. The efficacy and safety of different negative-pressure wound therapy gradients on flaps outcomes. Updates Surg. 2025 Dec;77(8):2643-2651. doi: 10.1007/s13304-025-02156-7. Epub 2025 Mar 23. PMID 40123035